CLINICAL TRIAL: NCT04943614
Title: Effect of BIODEX Balance System Training on Balance in Type II-diabetic Neuropathy.
Brief Title: Biodex Balance System Training in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00817 Rabia
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIODEX training group (Experimental): These individuals will receive conventional along with postural stability training with biodex balance system which stimulates specific movement patterns or strategies by placing markers on a specific location on-screen grid subject attempted to touch targets nine times using an onscreen cursor manoeuvred by the subject leg on the device platform
  Interventions: Other: Biodex balance system
- Conventional therapy group (Active Comparator): These individuals will perform balance exercises including proprioception exercises, balance board exercises, walking on different surfaces, Wobble board exercise and parallel bars for ambulatory training, range of motion exercises, foot care as a home program (advices).
  Interventions: Other: conventional exercises

INTERVENTIONS:
Other: Biodex balance system — BIODEX stability system (BIODEX Medical Systems Inc; Shirley, New York) offers a system that can deliver particular hip and ankle postural training strategy with external biofeedback as a monitor to enhance the reduced subclinical limitations of patients with diabetic neuropathy
  Arms: BIODEX training group
Other: conventional exercises — balance board exercises, walking on different surfaces, Wobble board exercise and parallel bars for ambulatory training, range of motion exercises, foot care as a home program. Same duration treatment
  Arms: Conventional therapy group

SUMMARY:
Type II-diabetic neuropathy is the most common and correlated problem with diabetes that deteriorates with the passage of time. Balance disorders are also resulting of movement strategy damage, biomechanical and mechanical disorientation. The balance disorder has been reported to be related to abnormal somatosensory feedback, which is utilized in the development of an interior depiction of body motion and position (inner model) in the central nervous system. The Biodex stability system offers a system that can deliver particular hip and ankle postural training strategy with external biofeedback as a monitor to enhance the reduced subclinical limitations of patients with diabetic neuropathy.

DETAILED DESCRIPTION:
Diabetes mellitus is one of the most common critical illnesses with a higher prevalence all over the world. Diabetic neuropathy is the most common and correlated problem with diabetes that deteriorates with the passage of time. Diabetic neuropathy is a progressive and complex disease, characterized by regular distal deterioration of peripheral nerves which lead to symptoms of sensory loss and pain. During normal situations, somatosensory inputs from the feet and legs participate in the stability of posture. Posture reflex and balance alignment are common findings in diabetic neuropathy because of reduced proprioception and rising time of reflex reactions. Balance disorders are also results of movement strategy damage, biomechanical and mechanical disorientation.

About 20-30% of patients with diabetic neuropathy suffer from neuropathic pains.

Neuropathic complications are prevalent among 39.6% of the diabetic population. Diabetic neuropathy lowers significantly the quality of life and considerably increases health expenses related to diabetes. Diabetic neuropathy patients exhibit stability disorders and are vulnerable to falls even with open eyes. The instability sources in patients with type-II diabetic neuropathy comprise the incapability of the central nervous system (CNS) to integrate properly available information of postural control and a shift of balance strategy from ankle-based to hip-based. Furthermore, a rise in the reliance on visual information and the use of vestibular information change the format of postural control in patients with diabetic neuropathy.

Stability can be referred to as the warmth of a dynamic system to different worries, and local constancy is the sensitivity of the structure to internal distresses, for example, natural fluxes like variation in muscle activity respond to gravity which occurs during stability. The impacts of such natural variations were inspected for assessing diverse measures of postural influence. Multiple studies on diabetic patients by neuropathic postural instability recommend relative shortfalls in their capability to sustain posture and specify higher instability as compared to non-diabetics and positive relations between falling and postural instability.

Moreover, studies of posture instability in diabetic patients with diabetic neuropathy have shown greater scores for postural stability indexes, area of sway, speed, greater ranges of the centre of pressure; increased values of the centre of mass variables and increase of sway power in less stable postures. Awareness and appropriately performing balance and stability training in patients involve comprehensive knowledge of the causes of postural complications. Postural control involves a composite organization that controls the equilibrium and orientation of the body during upright stand.

In addition, posture control involves multiple underlying physiological organizations and dependent upon six contexts: (a) cognitive processing, (b) sensory approaches, (c) movement approaches, (d) dynamics control (e), space orientation and (f) biomechanical task limitations. The sensory afferents sources which seem to participate in postural control comprise proprioception, visual systems, and vestibular. Subclinical and pathological constrictions in patients with diabetic neuropathy are because of context-specific and distinct instabilities like sensory and movement approaches. Reactive movement approaches are helpful for patients in developing multi-joint coordinated movement, and sensory approaches for selecting proper sensory information to control posture. The hip and ankle reactive movement approach reported being helpful to return the equilibrium of the body and keeping the feet in position. When people stand on a rigid surface, the ankle approach maintains balance with little movements in the form of an inverted pendulum. Rehabilitation and reactive movement strategies comprise the patient's exposure to external perturbations which differ in direction, amplitude, and speed. However, few studies have reported the correlation between balance training and external response. These trainings are useful to progress the sensory integration and dynamic balance capabilities of aged adults with a falling history and support for frail aged women in domestic care.

It also has been ideal to balance training at home. In addition, static-standing stability can be trained efficiently through weight-bearing exercise, and a visual guided weight-shifting drill can develop a standing balance mechanism of static balance in diabetic neuropathy patients. Like so, the BIODEX stability system offers a system that can deliver particular hip and ankle postural training strategy with external biofeedback as a monitor to enhance the reduced subclinical limitations of patients with diabetic neuropathy. As these patients are often of old age and have symptoms of instability identical to those of elder people, it is supposed that a balance-training platform with a BIODEX balance system may also improve balance in patients with diabetic neuropathy

ELIGIBILITY:
Inclusion Criteria:

* Age over 40 years both gender
* moderate & severe Type 2 diabetic neuropathy (modified Toronto Clinical Neuropathy Score) 9-11 = moderate neuropathy; ≥ 12 = severe neuropathy
* Ability to stand and walk independently.
* Berg balance score <50
* No cognitive impairments (Mini-Mental State Examination >23)

Exclusion Criteria:

* Individuals with other neurological deficits.
* Type 1 diabetic neuropathy.
* Diabetic ulcer, infection or partial amputation in feet.
* Orthopedic problem or severe pain affecting balance.
* History of repeated ankle sprains
* Visual problems.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | week 8
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete
Timed up and go test | week 8
  The Timed Up and Go (TUG) is a screening tool used to test basic mobility skills of frail elderly patients (60-90 years old). The TUG can be used with but is not limited to, persons with stroke.
  10s Completely independent With or without walking aid for ambulation and transfers
  < 20s Independent for main transfers With or without walking aid, independent for basic tub or shower transfers and able to climb most stairs and go outside alone
  > 30s Requires assistance Dependent in most activities
Functional reach test | week 8
  The Functional Reach Test is a single item test developed as a quick screen for balance problems in older adults.
  Interpretation: A score of 6 or less indicates a significant increased risk for falls. A score between 6-10 inches indicates a moderate risk for falls

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Afridi, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Armed Forces Institute of Rehabilitation And Medicine, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vinik AI, Nevoret ML, Casellini C, Parson H. Diabetic neuropathy. Endocrinol Metab Clin North Am. 2013 Dec;42(4):747-87. doi: 10.1016/j.ecl.2013.06.001. PMID 24286949
- [Background] Vincent AM, Callaghan BC, Smith AL, Feldman EL. Diabetic neuropathy: cellular mechanisms as therapeutic targets. Nat Rev Neurol. 2011 Sep 13;7(10):573-83. doi: 10.1038/nrneurol.2011.137. PMID 21912405
- [Background] Peltier A, Goutman SA, Callaghan BC. Painful diabetic neuropathy. BMJ. 2014 May 6;348:g1799. doi: 10.1136/bmj.g1799. PMID 24803311
- [Background] Abbott CA, Malik RA, van Ross ER, Kulkarni J, Boulton AJ. Prevalence and characteristics of painful diabetic neuropathy in a large community-based diabetic population in the U.K. Diabetes Care. 2011 Oct;34(10):2220-4. doi: 10.2337/dc11-1108. Epub 2011 Aug 18. PMID 21852677
- [Background] Akbari M, Jafari H, Moshashaee A, Forugh B. Do diabetic neuropathy patients benefit from balance training? J Rehabil Res Dev. 2012;49(2):333-8. doi: 10.1682/jrrd.2010.10.0197. PMID 22773533
- [Background] Pan X, Bai J. Balance training in the intervention of fall risk in elderly with diabetic peripheral neuropathy: A review. Int J Nurs Sci. 2014;1(4):441-5.
- [Background] Ghazal J, Malik AN, Amjad I. Task oriented training improves the balance outcome & reducing fall risk in diabetic population. Pak J Med Sci. 2016 Jul-Aug;32(4):983-7. doi: 10.12669/pjms.324.10092. PMID 27648053
- [Background] Singh R, Kishore L, Kaur N. Diabetic peripheral neuropathy: current perspective and future directions. Pharmacol Res. 2014 Feb;80:21-35. doi: 10.1016/j.phrs.2013.12.005. Epub 2013 Dec 25. PMID 24373831
- [Background] Schwenk M, Grewal GS, Holloway D, Muchna A, Garland L, Najafi B. Interactive Sensor-Based Balance Training in Older Cancer Patients with Chemotherapy-Induced Peripheral Neuropathy: A Randomized Controlled Trial. Gerontology. 2016;62(5):553-63. doi: 10.1159/000442253. Epub 2015 Dec 18. PMID 26678611